CLINICAL TRIAL: NCT04889326
Title: A Clinico-biological Database on Atypical Venous Thrombosis in the Context of anticovid19 Vaccination
Brief Title: Collection of the Thrombo-VaxCov Cohort
Acronym: THROMBO-VAXCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: ECH_2021_cb
Record Dates: First submitted 2021-04-27; First posted 2021-05-17 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Covid19; SARS-CoV Infection; Venous Thrombosis; Thrombocytopenia; Vaccination; Complications
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Venous Thrombosis; Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient hospitalized with atypical thrombosis within 4 weeks of anti-covid vaccination
  Interventions: Other: Retrospective data and biological samples

INTERVENTIONS:
Other: Retrospective data and biological samples — Analysis of data and biological samples collected during hospitalization:

SUMMARY:
In the context of anti-Covid19 vaccination, atypical thrombosis have occured and potential link with vaccination is under investigation.

This study collect clinical and biological data of all atypical thrombosis occurring within 4 weeks after antiCovid vaccination.

DETAILED DESCRIPTION:
In the context of anti-Covid19 vaccination, atypical thrombosis have occurred and potential links with vaccination is under investigation. In France, the study collect clinical and biological data of all atypical thrombosis occurring within 4 weeks after anti-Covid vaccination.

ELIGIBILITY:
Inclusion Criteria:

atypical thrombosis symptoms onset within 4 weeks of vaccination

Exclusion Criteria:

children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient hospitalized with atypical thrombosis occurring within 4 weeks of anticovid vaccination
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Functional outcome (modified rankin scale) | through study completion, an average of 1 years

SECONDARY OUTCOMES:
Recurrent vascular events | through study completion, an average of 1 years
Mortality | through study completion, an average of 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Cordonnier, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU lille, Lille, France

IPD SHARING:
Plan to Share IPD: Yes